CLINICAL TRIAL: NCT04126161
Title: HIP: Hip Imaging Protocol: the Comparison of Muscle Ultrasound-derived Parameters With CT Imaging-derived Parameters in Primary Total Hip Arthroplasty Patients.
Brief Title: HIP: Hip Imaging Protocol
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Mid-Study data analysis to determine if study should continue
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00102976
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Profiling Muscle
Keywords: muscle; ultrasound; CT; MuscleSound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CT (Active Comparator): Patients have standard of care CT prior to primary hip replacement
  Interventions: Procedure: CT
- Ultrasound (Experimental): Patients have ultrasound scans together with standard of care CT prior to primary hip replacement
  Interventions: Device: Ultrasound

INTERVENTIONS:
Procedure: CT — standard of care CT prior to primary hip replacement
  Arms: CT
Device: Ultrasound — Ultrasound scan together with standard of care CT prior to primary hip replacement
  Arms: Ultrasound

SUMMARY:
Objective measures of skeletal muscle features have previously been used to assess skeletal muscle quality. In certain clinical populations, such as intensive care (ICU) patients, specific features of the psoas muscle measured by abdominal CT have been used to assess the nutritional status of the patient. Abdominal CT is not performed routinely as it exposes the patient to ionizing radiation (X-rays) and can only be performed intermittently.

The measurement of the thigh muscles (rectus femoris muscle, part of the quadriceps muscle) by handheld musculoskeletal (MSK) ultrasound is a simple, safe (no ionizing radiation) and repeatable (can be easily performed on a daily basis) technique. A correlation has been shown between muscle parameters of the psoas muscle (abdominal CT) and the rectus femoris muscle (MSK). A direct comparison between muscle parameters of the same skeletal muscle measured with both CT and MSK has not been done.

Intramuscular adipose tissue (IMAT) is a measure of the extent of adipose tissue deposited within the muscle. It is a biomarker of muscle quality. The study objective is to compare muscle area and intramuscular adipose tissue (IMAT) content of rectus femoris muscle, measured by standard CT imaging with point of care handheld musculoskeletal (MSK) ultrasound in patients presenting for primary total hip arthroplasty. This patient group is chosen because they will have hip CT performed as standard of care prior to surgery.

DETAILED DESCRIPTION:
In our institution, all primary total hip arthroplasty patients receive abdominal CT that encompasses their hip as part of the standard clinical evaluation for hip surgery. This provides an opportunity to perform an MSK ultrasound at the same time.

Both CT and MSK have established imaging techniques of soft tissue. Both techniques provide a 2D digital slice representation. Although the image is black and white, there are a large number of intervals, up to 255, between the two extremes of black and white, termed grayscale. The application of an algorithm based upon the grayscale is used to define the different characteristics of the muscle, e.g. striated muscle versus fat infiltration. The algorithms used to measure muscle characteristics are entirely dependent on the originating imaging source. This means that an estimate of adipose using the CT algorithm is entirely independent of the algorithm applied to the MSK estimation of adipose.

This study, therefore, aims to determine how well the two imaging techniques correlate with each other when IMAT is measured by the two separate techniques.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip replacement

Exclusion Criteria:

* Revision hip replacement
* Ipsilateral knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
All IMAT | visit 1, up to 1 hour
  CT-derived area of intramuscular adipose tissue in cm2
%IMAT | visit 1, up to 1 hour
  Ultrasound-derived area of intramuscular adipose tissue in %

CONTACTS AND LOCATIONS:
Overall Officials: David MacLeod, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No